CLINICAL TRIAL: NCT00849940
Title: Validation of the CAS Medical System, Inc. FORE-SIGHT Near-Infrared Spectroscopy (NIRS) Monitor in Pediatric Subjects for Viscerosomatic Applications
Brief Title: Validation of Brain Oxygenation Monitor on Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: CAS Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00009391
Record Dates: First submitted 2009-01-22; First posted 2009-02-24 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cardiac Catheterization
Keywords: Spectroscopy; Near infrared; Oximetry; Hypoxemia; Tissue oxygenation; Pediatric
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAS NIRS FORE-SIGHT oximeter (Experimental): Pediatric patients presenting for cardiac catheterization.
  Interventions: Device: CAS NIRS FORE-SIGHT oximeter

INTERVENTIONS:
Device: CAS NIRS FORE-SIGHT oximeter — Comparison of non-invasive tissue oxygen saturation with blood sample-derived (calculated) tissue oxygen saturation.

SUMMARY:
The aim of this study is calibrate (adjust and tune) the CAS FORE-SIGHT Near-Infrared Spectroscopy (NIRS) monitor when used to measure the tissue oxygen saturation of internal organs (StO2). This is a measure of the amount of oxygen carried by the blood within the internal organs. In addition the study will assess the degree of similarities between StO2 and mean mixed venous oxygen saturation - a measure of the amount of oxygen carried in the blood returning to the heart.

DETAILED DESCRIPTION:
NIRS cerebral oximeters are FDA-approved devices used to measure oxygen saturation within the brain, in a similar manner to pulse oximeters that measure the oxygen saturation in the finger tip. The sensor pads are placed on the surface of the forehead and shine near-infrared light through the skull and brain tissue from which the brain tissue oxygen saturation is estimated. The same principles can be applied when the sensor pads are placed over the internal organs of the abdomen, for example, the liver. Currently the only way to accurately measure the oxygen saturation of internal organs is by the invasive placement of intravenous lines into the blood vessels of that organ. This study will determine if the NIRS sensors can reliably estimate the tissue oxygen saturation non-invasively by placing the pad over the skin of the abdomen.

The study will be conducted in pediatric patients who are undergoing cardiac catheterization, a procedure in which invasive lines are placed in order to get information about the heart. The procedure is always conducted under general anesthesia. During the cardiac catheterization procedure blood samples are routinely taken for oxygen saturation analysis. In the study two oximeter sensor pads will be placed on the forehead (one on each side) and two further oximeter sensor pads will be placed on the abdominal wall. The oxygen saturation values from all oximeter sensors will be recorded continuously throughout the cardiac catheterization procedure and will be compared to the oxygen saturation values from the blood samples. In addition to the routine blood samples taken as part of the cardiac catheterization, one blood sample will be taken when the invasive line is within the right hepatic (liver) vein.

The information from this study will determine how well the oximeter sensors estimate the oxygen saturation of both the internal organs (StO2) and the blood returning to the heart (mean mixed venous oxygen saturation).

ELIGIBILITY:
Inclusion Criteria:

* ≤ 18 years old
* ≥ 2.5 kg and ≤ 40 kg weight
* Undergoing cardiac catheterization at Duke pediatric cardiac catheterization laboratory

Exclusion Criteria:

* Known structural neurologic or craniofacial disease
* Arterial catheter placement not part of planned catheterization procedure
* Anemia (hemoglobin < 10 g/dl)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2009-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, FCRA, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Started | 72
Completed | 68
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 72
  Between 18 and 65 years | 0
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 34
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 66
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of NIRS Sensor to Estimate Flank Tissue Oxygen Saturation
Description: The flank tissue oxygen saturation (%) is determined from simultaneous arterial and venous blood samples processed through a blood gas machine. The blood oxygen saturation of the samples are entered into an equation to yield the best estimate of flank tissue oxygen saturation. This value is then compared to the NIRS oxygen saturation (%) displayed on the monitor. Accuracy is used to describe how close the NIRS oxygen saturation is to the flank tissue oxygen saturation. It can be expressed in terms of shots on target: bias (%) = how close are the shots to the bulls eye and precision (%) is how close are the shots to each other.
  oxygen saturation when measured displayed NIRS value of the tissue sensor placed over the flank to a reference CO-oximetry model, reported as bias and precision. The model is weighted as 30:70 arterial: central venous oxygen saturation when measured by blood gas co-oximetry.
Time Frame: Data collected from individual participants over 4 hour timeframe.
Population: Weight range 3.9 - 49.5 kg; age 0.2 - 12.3 years represent the values of the participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 43
percentage of oxygen saturation | -0.67 (4.88)

2. Primary Outcome: Accuracy of NIRS Sensor to Estimate Intestine Tissue Oxygen Saturation
Description: The intestine tissue oxygen saturation (%) is determined from simultaneous arterial and venous blood samples processed through a blood gas machine. The blood oxygen saturation of the samples are entered into an equation to yield the best estimate of intestine tissue oxygen saturation. This value is then compared to the NIRS oxygen saturation (%) displayed on the monitor. Accuracy is used to describe how close the NIRS oxygen saturation is to the intestine tissue oxygen saturation. It can be expressed in terms of shots on target: bias (%) = how close are the shots to the bulls eye and precision (%) is how close are the shots to each other.
Time Frame: Data collected from individual participants over 4 hour timeframe.
Population: Weight 2.9 - 24.0 kg; age 0.04 - 9.8 years represent the values of the participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 45
percentage of oxygen saturation | 1.57 (4.41)

3. Primary Outcome: Accuracy of NIRS Sensor to Estimate Hepatic Tissue Oxygen Saturation
Description: The hepatic tissue oxygen saturation (%) is determined from simultaneous arterial and venous blood samples processed through a blood gas machine. The blood oxygen saturation of the samples are entered into an equation to yield the best estimate of hepatic tissue oxygen saturation. This value is then compared to the NIRS oxygen saturation (%) displayed on the monitor. Accuracy is used to describe how close the NIRS oxygen saturation is to the hepatic tissue oxygen saturation. It can be expressed in terms of shots on target: bias (%) = how close are the shots to the bulls eye and precision (%) is how close are the shots to each other.
Time Frame: Data collected from individual participants over 4 hour timeframe.
Population: Weight 2.9 - 25.4 kg; age 0.04 - 10.2 years represent the values of the participants analyzed.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 63
percentage of oxygen saturation | 0.04 (5.63)

4. Secondary Outcome: Correlation Between Somatic StO2 and Cerebral SctO2 Oxygen Saturation
Time Frame: Data collected from individual participants over 4 hour timeframe
Population: Data not collected
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation Between NIRS Derived Estimate of Hemoglobin Concentration and Measured Arterial Blood Hemoglobin Concentration.
Time Frame: Data collected from individual participants over 4 hour timeframe
Population: Data not collected.
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CAS NIRS FORE-SIGHT Oximeter
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 0/72

LIMITATIONS AND CAVEATS:
Blood samples collected from pediatric patients undergoing cardiac catheterization. Venous blood samples taken from within IVC as close to the tissue of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes